CLINICAL TRIAL: NCT05886361
Title: Somatic Symptoms in Autism Spectrum Disorder: Data Integration
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202206027RINA
Record Dates: First submitted 2023-05-04; First posted 2023-06-02 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2022-06

CONDITIONS: Autism Spectrum Disorder; Somatic Symptom Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- ASD: Diagnosed with DSM-5 autism spectrum disorder
  Interventions: Other: No intervention involved
- Clinical: Patients with anxiety, depression, somatic symptoms which are non-psychotic and non-organic
  Interventions: Other: No intervention involved
- Control: Healthy control without psychiatric disorder or chronic somatic symptoms
  Interventions: Other: No intervention involved

INTERVENTIONS:
Other: No intervention involved — No intervention involved

SUMMARY:
Autistic patients have higher chances commorbid somatic symptoms. Therefore, it leads to more health-related concerns, such as autoimmune disease, gastrointestinal disease, cardiovascular disease, autonomic disorders. On average, autistic patient's life span is 16 years shorter than non-autistic patients. Furthermore, autistic patients are not able to convey or communicate their somatic symptoms in a clear and comprehensive manner. This leads to unable to receive proper health care in a timely manner.

ELIGIBILITY:
Inclusion Criteria:

* ASD group: diagnosed with DSM-5 autism spectrum disorder
* clinical group: anxiety, depression, somatic disorder who are non-psychotic and non-organic
* control group: healthy control without psychiatric disorder or chronic somatic symptoms
* age between 15 and 70

Exclusion Criteria:

* psychiatric disorders such as schezophrenia, mood disorder.
* major physical disorder which can be potentially lethal
* who cannot read or comprehend the survey and questionnaire

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: as mentioned earlier, it is a retrospective study with existed data. Therefore, the 1423 participants are already collected in the past. We separate these existed data into three groups as mentioned in the eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 1423 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Patient health questionnaire-15, PHQ-15 | 8 years
  range from 0 to 2 for each item, total score range from 0 to 30. Higher the score, worse the level of somatization
Health assessment questionnairse, HAQ | 8 years
  range from 0 to 3 for each item. Higher the score, worse the disability
Beck depression inventory, BDI | 8 years
  range from 0 to 3 for each item. Higher the score, worse the depression
Beck anxiety inventory | 8 years
  range from 0 to 3 for each item. Total score 0 to 63. Higher the score, worse the anxiety